CLINICAL TRIAL: NCT07328503
Title: A Phase II Study to Examine the Impact of CD22 CAR T-cells to Extend the Duration of Remission Following Commercial CD19 CAR T-cells in Children, Adolescents, and Adults With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: CD22 CAR T-cells to Extend Remission Following Commercial CD19 CAR T-cells in Children, Adolescents, and Adults With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001986; 001986-C
Record Dates: First submitted 2026-01-08; First posted 2026-01-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-12

CONDITIONS: Acute Lymphoblastic Leukemia; B-All
Keywords: B-All; Acute Lymphoblastic Leukemia; CD-22 Expressing Tumor; CD-19 expressing tumor; Adoptive Immunotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Lymphodepleting chemotherapy followed by CD22 CAR T-cells
  Interventions: Biological: CD22 CAR-transduced T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CD22 CAR-transduced T cells — CD22-CAR-transduced T cells on D0 after lymphodepleting preparative regimen
Drug: Cyclophosphamide — Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the patient s body weight, at 500 mg/m^2/dose after fludarabine infusion on days -3 and -2.
Drug: Fludarabine — Fludarabine is administered as an IV infusion in an appropriate solution over 30 minutes on days -5 through -2. To prevent undue toxicity the dose will be based on BSA (30 mg/m^2/dose).

SUMMARY:
Background:

Acute lymphoblastic leukemia (ALL) is a type of blood cancer. Chimeric antigen receptor (CAR) therapy involves taking immune cells (T cells) from a person and modifying them to better target cancer cells. CAR T-cell therapy that targets a marker called CD19 has been show to can cure ALL in many children and adults. But in about 50% of patients, the ALL comes back within a year. Researchers want to find out if a second treatment with CAR T-cell therapy that targets a different marker, CD22, can keep the cancer away longer.

Objective:

To see if CD22 CAR T-cell therapy can keep ALL away longer.

Eligibility:

People aged 3 to 65 years who have no signs of cancer after CD19 CAR T-cell treatment for ALL.

Design:

Participants will be screened. They will have imaging scans and tests of their heart function. A sample of tissue (biopsy) will be collected from their bone marrow. They will have a fluid sample collected from the area around their spinal cord.

Participants will undergo collection of their white blood cells (T cells) during a procedure called leukapheresis. Blood will be taken from their body through a vein. The blood will pass through a machine that separates out the T cells. The remaining blood will be returned to the body through a different vein. The cells will be altered in a lab to create CD22 CAR T-cell therapy.

Participants will take drugs over 4 consecutive days to prepare their body for the CAR T-cell therapy; then they will receive their modified T cells through a tube inserted into a vein. Some people may need to stay in the hospital during treatment.

Participants will have follow-up visits for 2 years.

DETAILED DESCRIPTION:
Background:

* Despite impressive cure rates in children and young adults with B-cell acute lymphoblastic leukemia (B-ALL) generally, patients with relapsed/refractory disease have historically suffered from limited treatment options. CD19 and CD22 chimeric antigen receptor (CAR) T-cells are effective at inducing remission in the majority of children and young adults with relapsed/refractory B-ALL.
* However, remissions are often not durable, and many patients will relapse in the absence of a consolidative hematopoietic stem cell transplant (HSCT), which is associated with high morbidity and mortality.
* Leukemic antigen escape has led to the interest in multi-antigen targeting approaches, targeting both CD19 and CD22 to enhance the long-term effectiveness of CAR T-cells. We have previously treated patients on phase 1/2 clinical trials using a bivalent CD19/22 CAR T-cell as well as a bicistronic CD19xCD22 CAR T-cell as combinatorial strategies.
* Some of the best long-term results in the literature have been seen with co-infusion of CD19 and CD22 CAR T-cells. Two FDA-approved CD19 CAR T-cell products are available commercially, and our phase 1/2 trial of CD22 CAR T-cells has demonstrated efficacy and safety.
* The use of CD22 CAR T-cells as consolidation of CD19 CAR T-cell-induced remission offers the potential to extend the durability of remission while limiting the toxicity associated with HSCT.

Objective:

-To determine the 1-year relapse-free survival (RFS) from the time of CD22 CAR T-cell infusion.

Eligibility:

-Participants aged 3-65 years who have relapsed/refractory B-ALL with a history of demonstrated expression of CD19 and CD22 and have achieved an MRD-negative remission after receiving an FDA-approved CD19 CAR T-cell product.

Design:

* Single-arm study with 4 days lymphodepleting preparative regimen, including fludarabine and cyclophosphamide, followed by CD22 CAR T-cells administration.
* Participants will be evaluated for toxicity, antitumor effects, CAR expansion and persistence, and other biological correlatives for 2 years after cell infusion.
* The trial will accrue 16 evaluable participants. The accrual ceiling for the trial is 20 participants to account for inevaluable participant and screen failures.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have documentation of pathologic confirmation of a diagnosis of relapsed/refractory B cell acute lymphoblastic leukemia (ALL).
* History of CD19 and CD22 expression on malignant cells at diagnosis or relapse.
* Age between >= 3 years and <= 65 years
* Participants must have received an FDA-approved CD19 CAR T-cell construct for treatment of B cell ALL within the time period of >= 2 months and <= 7 months prior to apheresis or lymphodepleting (LD) (if apheresis is not done on this protocol).
* Must be in an MRD-negative remission as demonstrated by flow cytometry at screening.
* Must be ineligible for or unwilling to undergo allogeneic stem cell transplant (SCT).
* Clinical performance status (PS): Karnofsky >= 50% (participants >= 16 years of age), or Lansky scale >= 50% (participants < 16 years of age). Participants who are unable to walk because of paralysis, but who are upright in a wheelchair may be considered eligible.
* Must have no ongoing signs of CRS from prior CAR T cell infusion and/or ICANs at screening.
* Participants must have adequate organ function as defined below:

  * Total bilirubin <= 2 x institutional upper limit of normal (ULN)
  * Aspartate Aminotransferase (AST) <= 10 x ULN
  * Alanine Aminotransferase (ALT) <= 10 x ULN
  * creatinine <= the maximum for age listed below OR measured creatinine clearance >= 60 mL/min/1.73 m^2 for participants with

creatinine levels above the max

* Age: <=5, Maximum Serum, Creatinine <= .8 mg/dL
* Age: >5 to <=10, Maximum Serum, Creatinine <= 1.0mg/dL
* Age: >10, Maximum Serum, Creatinine <= 1.2mg/dL

  * A participant may have continued to expect CAR T cell-associated cytopenias of any grade.
  * Cardiac function: left ventricular ejection fraction>= 45% or fractional shortening >= 28%.
  * Pulmonary function: baseline oxygen saturation >= 92% on room air; participants with respiratory symptoms (e.g., dyspnea, hypoxia <92%) must have a diffusing capacity of the lungs for carbon monoxide (DLCO)/adjusted > 45%.
  * Women of childbearing potential (WOCBP) must agree to use highly effective contraception (hormonal, intrauterine device (IUD), abstinence, surgical sterilization) at the study entry and up to 12 months after the last dose of combined chemotherapy.

Note: WOCBP is defined as any individual who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

Men able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and up to 7 months after the last dose of study drugs. We also will recommend men ask their partners to be on highly effective birth control (hormonal, IUD, surgical sterilization). Individuals able to father a child must not freeze or donate sperm within the same period.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 6 months after the last dose of the study drug(s).
* Participants must be enrolled on protocol 15-C-0028, Follow-Up Evaluation for Gene- Therapy Related Delayed Adverse Events after Participation in Pediatric Oncology Branch Clinical Trials.
* Ability of participant or /Legally Authorized Representative (LAR) to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Any central nervous system (CNS) involvement or signs of non-CNS extramedullary disease.
* Any active graft versus host disease (GVHD) in participants who are post-HSCT.
* Participants with disease recurrence requiring therapy post CD19 CAR. Note: Maintenance therapy post CD19 CAR (e.g., vincristine or tyrosine kinase inhibitor) for remission maintenance is allowed and will require a 1-week washout prior to apheresis or LD (if apheresis is not done on this protocol).
* Any investigational agent within 1 week before apheresis or LD (if apheresis is not done on this protocol).
* Pregnancy confirmed with beta-human chorionic gonadotropin (beta-HCG) serum or urine test performed at screening.
* Human immunodeficiency virus (HIV) infection, as measured by seropositivity for (HIV) antibody.
* Hepatitis B virus (HBV) infection, as measured by positivity for hepatitis B surface antigen (HBsAg).
* Hepatitis C virus (HCV) infection, as measured by seropositivity for hepatitis C.
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biological composition to any agent used in the study or in the manufacturing of cells.
* Uncontrolled, symptomatic intercurrent illness evaluated by medical history, physical exam, and/or laboratory testing, or social situation that would limit compliance with study requirements or would pose an unacceptable risk to the participant.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
1-year RFS (recurrence free survival) | 1 year post cell infusion
  RFS of participants will be assessed by a Kaplan-Meier curve. The RFS probability and the median RFS will be reported along with 95% confidence intervals.

SECONDARY OUTCOMES:
2-year RFS | 2 years post cell infusion
  RFS probability will be reported along with 95% confidence intervals.
1-year and 2-year OS (overall survival) | 2 years post cell infusion
  OS of participants will be assessed by Kaplan-Meier curves along with 95% confidence intervals. OS will be described for participants with HSCT and without HSCT, for descriptive purposes, along with 95% confidence intervals.
Short-term safety | 28 days post cell infusion
  Short-term safety of CD22 CAR T-cell infusion for participants in remission after CD19 CAR T-cell infusion will be evaluated by describing: CRS incidence and severity per ASTCT; ICANS incidence and severity per ASTCT; EC-HS incidence and severity; ICAHT incidence and severity; and incidence of grade >= 3 serious adverse events per CTCAE v.5.0.
Long-term safety | up to 2 years post cell infusion
  Long-term safety of CD22 CAR T-cell infusion for participants in remission after CD19 CAR T-cell infusion will be evaluated by describing: incidence of severe adverse events related to CD22 CAR T-cells
RFS from the time of additional CD22 CAR T-cell infusions | up to 2 years post-cell infusion
  RFS probability will be reported along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Silbert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001986-C.html